CLINICAL TRIAL: NCT00410033
Title: Safety/Efficacy Trial Using Stored Serum Samples to Investigate the Immunogenicity of Insulin Aspart and Soluble Human Insulin in Children and Adolescents From Onset of Type 1 Diabetes
Brief Title: Comparison of Antibody Levels in Children and Adolescents After Initiation of Insulin Therapy by Either Insulin Aspart or Soluble Human Insulin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANA-1676
Record Dates: First submitted 2006-12-11; First posted 2006-12-12 (Estimated); Last update posted 2016-12-22 (Estimated); Status verified 2016-12

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — Insulin, Isophane; Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: soluble human insulin
Drug: isophane human insulin
Drug: insulin aspart

SUMMARY:
This trial is conducted in Europe. This is a single-centre, retrospective trial aiming at comparing the antibody levels in children and adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any trial-related activities
* Any subjects at onset of Type 1 Diabetes
* Treatment with either Insulin Aspart and Soluble Human Insulin or Soluble Human Insulin and Isophane Human Insulin / Mixtard® for at least 9 months from the time of diagnosis of diabetes

Exclusion Criteria:

* Treatment with immunosuppressive agents
* For the Insulin Aspart + Isophane Human Insulin: Treatment with insulin analogues other than Insulin Aspart or treatment with fast acting human insulin for a period of 7 days or more during the treatment period
* For the Soluble Human Insulin and Isophane Human Insulin group: Treatment with insulin analogues
* Other diseases influencing immune response
* Unable or unwilling to provide consent

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 74 (Actual)
Dates: Start 1989-12; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Insulin aspart specific, human insulin specific and cross reacting antibodies | measured up to at most 2.5 years after diagnosis

SECONDARY OUTCOMES:
HbA1c
Insulin requirements
Incidence of hypoglycaemic episodes

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Linköping, Sweden

REFERENCES:
- [Result] Holmberg H, Mersebach H, Kanc K, Ludvigsson J; Insulin Aspart Study Group on Immunogenicity. Antibody response to insulin in children and adolescents with newly diagnosed Type 1 diabetes. Diabet Med. 2008 Jul;25(7):792-7. doi: 10.1111/j.1464-5491.2008.02468.x. PMID 18644065
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com